CLINICAL TRIAL: NCT00349856
Title: Dispensing Overnight Study in Lenses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Cooper Companies (Industry)
Responsible Party: Craig Woods, Research Manager, Centre for Contact Lens Research
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: P/209/04/O
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator)
  Interventions: Device: Biofinity

INTERVENTIONS:
Device: Biofinity — Soft contact lens
  Other Names: Purevision

SUMMARY:
The purpose of the study is to evaluate the fit and performance of an investigational soft contact lens in comparison with a currently marketed lens. Both lenses will be worn on a continuous wear basis, which means the lenses will be worn while sleeping.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the fit and performance of an investigational soft contact lens in comparison with a currently marketed lens. Both lenses will be worn on a continuous wear basis, which means the lenses will be worn while sleeping. Physiological changes will be monitored and subjective ratings collected.

ELIGIBILITY:
Inclusion Criteria:

1. Has had an oculo-visual examination in the last 2 years.
2. Is between 18-45 years old and has full legal capacity to volunteer.
3. Has read and understood the Information Consent Letter
4. Is willing and able to follow participant instructions for product usage and meet the protocol-specified schedule of follow-up visits.
5. Is correctable with the prescription of the available lenses (-1.00 to -4.00 DS in 0.50D step).
6. Is correctable to at least 20/40 distance visual acuity with contact lenses in each eye.
7. Is a current soft contact lens wearer (both daily wear and extended wear experience allowed).
8. Has refractive astigmatism of <= 1.00 diopters
9. Has clear corneas and ocular clinical findings considered to be "normal".

Exclusion Criteria:

1. Has any systemic disease affecting ocular health.
2. Is using any systemic or topical medications that will affect ocular health.
3. Has any ocular pathology or severe insufficiency of lacrimal secretion (dry eyes) that would affect the wearing of contact lenses.
4. Has any clinically significant lid or conjunctival abnormalities, neovascularization, corneal scars or corneal opacities.
5. Has limbal injection, bulbar injection or corneal staining that, in the Investigator's opinion, is clinically significant.
6. Has never worn contact lenses before.
7. Has corneal distortion resulting from rigid lens wear.
8. Is aphakic.
9. Has undergone corneal refractive surgery.
10. Is participating in any other type of clinical or research study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this trial is to assess safety of the investigational | study visits, three monthly

SECONDARY OUTCOMES:
The secondary objective of this trial is to assess the subjective responses to comfort with both the investigational and marketed lenses. | study visits, three monthly

CONTACTS AND LOCATIONS:
Overall Officials: Desmond Fonn, MOptom, Principal Investigator — Centre for Contact Lens Research, University of Waterloo.
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada